CLINICAL TRIAL: NCT04894838
Title: DIStal gastriC Bypass OUtcome in Revision SurgEry After Roux-en-y Gastric Bypass
Acronym: DISCOURSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, M.J. Wiezer, Dr. M.J. Wiezer, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL75322.100.20/R20.093
Record Dates: First submitted 2021-04-13; First posted 2021-05-20 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Obesity, Morbid; Weight Gain
Keywords: Obesity; Weight regain; Failed RYGB; Distal gastric bypass
MeSH Terms: conditions — Obesity, Morbid; Weight Gain; Obesity

STUDY DESIGN:
Intervention Model Description: In total, 150 morbidly obese patients are eligible for distalisation surgery following RYGB. The participants will be randomised into DGB type I (group a) or DGB type II (group b). The study population consists of morbidly obese patients with insufficient weight loss or weight regain following primary Roux-en-Y gastric bypass, who are eligible for distalisation surgery.
Who Masked: Participant
Masking Description: Patients who meet the eligibility criteria will be included in this trial at the outpatient clinic of the participating bariatric centres after informed consent is obtained. The participating patients will be randomised into one of the surgical techniques: type I or type II DGB. Randomisation will take place in the operating room through an internet-based randomisation system in REDCap. Only the participants are blinded to the treatment allocation. The randomisation table will be created by an independent epidemiologist in the St. Antonius hospital, ensuring concealment of treatment allocation. Participants will be randomised in equal numbers to both interventions. The randomisation will be stratified by participating hospitals to ensure participants are evenly allocated to each treatment arm at each participation hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal gastric bypass type I (Experimental): Laparoscopic distalisation of RYGB type I. The RYGB is modified by dividing the Roux limb (AL) at the jejuno-jejunal anastomosis and re-anastomosed distally to 200 cm from the ileocecal valve using linear staplers, creating a long biliopancreatic limb (BPL). In cases of initial AL lengths shorter than 100 cm, the CC lengths should be adjusted to create a TALL of at least 300 cm.
  Interventions: Procedure: Distal gastric bypass
- Distal gastric bypass type II (Experimental): Laparoscopic distalisation of RYGB type II. The RYGB is modified by dividing the BPL at the jejuno-jejunal anastomosis and re-anastomosed distally to 200 cm from the ileocecal valve using linear staplers, creating a long AL.
  Interventions: Procedure: Distal gastric bypass

INTERVENTIONS:
Procedure: Distal gastric bypass — Distal gastric bypass, revisonal surgery after failed RYGB

SUMMARY:
This study is designed as a prospective multicenter randomized controlled clinical trial comparing two surgical techniques of distal gastric bypass (DGB) in revisional surgery following failed Roux-en-Y gastric bypass. Patients will be randomly allocated 1:1 to A) DGB with lengthening of the BPL (DGB type I) or B) DGB with extended AL (DGB type II). Randomisation is stratified for participating center. The study will be performed in a clinical and out-patient setting with regular visits at 1.5, 3, 6, 12, 18, 24 and 36 months post intervention. The study will be set up as a multicenter study with bariatric centers: St. Antonius hospital, Groene Hart hospital, OLVG, Rijnstate hospital, Elisabeth Twee-steden Hospital, Bravis hospital, Medisch Centrum Leeuwarden, Catharina Hospital.

DETAILED DESCRIPTION:
Rationale: Up to 35% of morbidly obese patients undergoing Roux-en-Y gastric bypass (RYGB) fail to lose sufficient weight or regain excessive weight after initial weight loss. Currently, there is no standardized approach to revisional surgery after failed RYGB. Distalisation of the RYGB limbs (DGB), with shortening of the common channel and extending either the alimentary limb (AL) or biliopancreatic limb (BPL), can be performed as revisional surgery to induce additional weight loss. To date, there is no general consensus as to optimal surgical technique or limb lengths to be used in distalisation of RYGB in both literature as well as clinical practice.

Objective: The aim of this study is to investigate the effect of two distalisation techniques of a gastric bypass in revisional surgery with standardised limb lengths in total weight loss (TWL) and the need for treatment for protein calorie malnutrition (PCM). In this randomised controlled trial DGB with lengthening of the BPL (DGB type I) will be compared to DGB with extended AL (DGB type II) in order to conclude which surgical technique is the optimal therapeutic strategy as revision surgery following Roux-en-Y gastric bypass.

Study design: A multicentre randomised controlled trial.

Study population: Morbidly obese patients with insufficient weight loss or weight regain following primary RYGB, who are eligible for distalisation surgery.

Intervention: A total of 150 participants will be randomised over two treatment groups: group A will undergo DGB type I and group B will undergo DGB type II.

Main study endpoints: Primary endpoints: %TWL 1 year after treatment and need for treatment of PCM. Secondary endpoints: weight loss, co-morbidity remission, PCM grading (debilitating defecation patterns, temporary total parenteral nutrition treatment, revision, mortality), morbidity, nutritional deficiencies, quality of life and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years;
* BMI ≥40 kg/m2 or BMI ≥35 kg/m2 with obesity related comorbidity;
* Weight regain or insufficient weight loss (EWL<50% or TWL<20%)15,16 following RYGB;
* Multidisciplinary team screening at one of the bariatric centres;
* Informed consent and willing to enter the follow-up program.

Exclusion Criteria:

* Failed Roux-en-Y gastric bypass due to anatomic, surgical reasons (gastric pouch dilatation >50 mL, gastro-gastric fistula, gastro-jejunostomy);
* Distalisation of RYGB is technical infeasible (judgment by surgeon);
* Inflammatory bowel disease, celiac disease, irritable bowel syndrome and other causes of chronic diarrhea;
* Severe concomitant disease (such as carcinomas and neurodegenerative disorders);
* Pregnant women;
* Noncompliance in follow-up or unwilling to undergo surgery;
* Inability of reading/understanding and filling out questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 1 year post-operative
  Percentage total weight loss (%TWL) 1 year after treatment
Number of Participants with development of protein calorie malnutrition (PCM) | 1 year postoperative
  >6 times/day defecation patterns with diarrhea, assessed by fecal score questionnaire

SECONDARY OUTCOMES:
Weight loss | Up to 3 year follow up
  Patient weight in kilograms is collected preoperative up to 3 years follow-up to determine weight loss.
TWL | 3, 6, 12, 18, 24, 36 month follow up
  Weight loss in kilograms at a follow-up time point divided by weight in kilograms measured at DGB
Defecation pattern | 3, 12 and 36 months postoperative
  Faecal score questionnaire to measure defecation frequencey and consistency
PCM grading | up to 3 year follow up
  Information is collected about each patient who has undergone DGB to ascertain debilitating defecation patterns (grade I), requirement of f participants requiring temporary total parenteral nutrition (grade II, revision surgery (grade III), and mortality (grade IV) after DGB.
Complications | uo to 3 year follow up
  Information is collecting regarding the occurrence of one or more defined adverse events following DGB. Defined adverse events collected are: unplanned readmission to hospital, unplanned admission to the intensive care unit, unplanned return to the operating theatre, prolonged length of stay in hospital, and death. The reason for any of the events is also collected. If death occurs, the cause of death is collected to determine the likelihood of the death being caused by the DGB.
Quality of life questionnaire | 3, 12 and 36 months postoperative
  BODY-Q questionnaire
Impact defecation pattern questionnaire | 3, 12 and 36 months postoperative
  Fecal incontinence quality of life scale FIQL questionnaires
Patient satisfaction questionnaire | 1 and 3 year postoperative
  Self-designed 5-point scale measuring instrument for patient satisfaction
Eating behaviour questionnaire | 3, 12 and 36 months postoperative
  Three factor earing questionnaire TFEQ R21

CONTACTS AND LOCATIONS:
Overall Officials: M.J. Wiezer, PhD, MD, Principal Investigator — St. Antonius Hospital
Locations (8):
- Netherlands (8):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Bravis Hospital, Roosendaal, North Brabant
  - Elisabeth-Tweesteden Hospital, Tilburg, North Brabant
  - OLVG, Amsterdam, North Holland
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Groene Hart Hospital, Gouda, South Holland
  - St. Antonius hospital, Nieuwegein, Utrecht

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT04894838/Prot_SAP_000.pdf